CLINICAL TRIAL: NCT03743311
Title: The Russian Multicenter Observational Program Obtaining of Data on the Impact of Different Treatment Modalities on the Quality of Life of the Patients With Acute and Chronic Hemorrhoid Disease
Brief Title: Data on the Impact of Different Treatment on the Quality of Life of Patients With Acute and Chronic Hemorrhoid Disease
Acronym: EQUALISER
Status: Completed | Type: Observational
Sponsor: Servier Russia (Industry)
Responsible Party: Sponsor
Other Study IDs: IC4 -05682-058-RUS
Record Dates: First submitted 2018-11-13; First posted 2018-11-16 (Actual); Results first posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Hemorrhoids
MeSH Terms: conditions — Hemorrhoids | interventions — Hemorrhoidectomy; Thrombectomy; S 5682; Psychotherapy, Multiple

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Surgical treatment of Hemmorhoid: Patients after surgical treatment (Instrumental Invasive Surgical Procedures or Thrombectomy, Hemorrhoidectomy etc.)
  Interventions: Procedure: Hemorrhoidectomy, Thrombectomy , Operation on Longo method
- Conservative treatment of Hemmorhoid: Patients taken conservative treatment (Detralex)
  Interventions: Drug: Detralex
- Combined treatment of Hemmorhoid: Combined treatment patients (surgery and conservative treatment)
  Interventions: Other: Combined therapy

INTERVENTIONS:
Procedure: Hemorrhoidectomy, Thrombectomy , Operation on Longo method — Surgical procedures for treatment of Hemorhoid
  Groups: Surgical treatment of Hemmorhoid
Drug: Detralex — Conservative treatment of Hemorhoid
  Groups: Conservative treatment of Hemmorhoid
Other: Combined therapy — Surgical + conservative treatment of Hemorhoid
  Groups: Combined treatment of Hemmorhoid

SUMMARY:
The program is aimed at obtaining data on the impact of the method and type of treatment on the quality of life of patients with acute or chronic hemorrhoids with option of conservative treatment with Detralex

DETAILED DESCRIPTION:
Changes in the quality of life of patients suffering from acute or chronic hemorrhoids within 1 month after presenting to a doctor, in general population and in specific demographic and clinical groups.

The program included patients who presented to a doctor for acute or chronic hemorrhoids. All the treatment was fully compliant with the conventional clinical practice, instructions for medical use of drugs and a specific clinical situation. The standard parameters usually evaluated in patients with hemorrhoids were studied during the program. In addition, at the first visit to the doctor and at the end of the study, the patient filled out an SF-36 questionnaire for assessing the QoL

The general population of patients included in the program, the following three groups of patients were considered:

* Group 1, with only conservative (medical) therapy during the study;
* Group 2, with conservative (medical) therapy and additional minimally invasive procedure during the study (no surgery);
* Group 3, with conservative (medical) therapy and additional surgery for hemorrhoids during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years;
2. Providing written information to a patient about inclusion in the program, and his/her consent to participate in it,
3. Absence of conditions requiring urgent medical care and not related to hemorrhoids;
4. The patient was diagnosed with:

   * Acute hemorrhoids;
   * Exacerbation of chronic hemorrhoids;
   * Chronic hemorrhoids

Exclusion Criteria:

1. The patient is consulting for an urgent issue not related to hemorrhoids;
2. The presence of severe systemic diseases;
3. Pregnancy;
4. Inability to understand the meaning of the Program and follow the doctor's recommendations
5. Patients with inflammatory bowel diseases
6. Patients with concomitant diseases of the anal canal
7. Patients taking anticoagulants;
8. Patients with previous anorectal surgeries, including hemorrhoidectomy or excision of anal fistula.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute or chronic hemorrhoids.
Sampling Method: Non-Probability Sample
Enrollment: 1032 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olga LINNIK, Study Chair
Locations (1):
- Pirogov National Surgery Center, Moscow, Pervomaisrfya 70, Russia

REFERENCES:
- Available data/document: the SF36 scale questioner — https://clinmedjournals.org/articles/jmdt/jmdt-2-023-figure-1.pdf — The scale the SF36 scale questioner can be sent by email.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Conservative Treatment of Hemmorhoid | Combined Treatment of Hemmorhoid | Surgical Treatment of Hemmorhoid
Started | 311 | 298 | 423
Completed | 311 | 298 | 423
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conservative Treatment of Hemmorhoid | Combined Treatment of Hemmorhoid | Surgical Treatment of Hemmorhoid | Total
Number analyzed (Participants) | 311 | 298 | 423 | 1032
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 289 | 274 | 396 | 959
  >=65 years | 22 | 24 | 27 | 73
Age, Continuous [Mean (Full Range); unit: years] | 42.9 [18 to 90] | 44.2 [19 to 78] | 46.9 [20 to 94] | 44.9 [18 to 94]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: There is no data about sex of 2 participants in Group 1 There is no data about sex of 3 participants in Group 3
  Participants
    number analyzed (Participants) | 309 | 298 | 420 | 1027
    Female | 171 | 139 | 209 | 519
    Male | 138 | 159 | 211 | 508
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 311 | 298 | 423 | 1032
patients with acute or chronic hemorrhoids [Count of Participants; unit: Participants] | 311 | 298 | 423 | 1032

OUTCOME MEASURES:

1. Primary Outcome: Changes in the Quality of Life of Patients Suffering From Acute or Chronic Hemorrhoids Within 1 Month After Presenting to a Doctor (Visit V0 vs Visit3)
Description: The Short Form (36) Health Survey (SF36 ) scale questioner was used. SF36 is is a 36-item, patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Time Frame: 1 month after presenting to a doctor
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Surgical Treatment of Hemmorhoid | Conservative Treatment of Hemmorhoid | Combined Treatment of Hemmorhoid
Number analyzed (Participants) | 311 | 298 | 423
units on a scale
  Physical functioning | 16.5 [3.4 to 29.6] | 11.1 [2.7 to 19.5] | 13.7 [6.4 to 21]
  Role physical | 15.5 [10 to 21] | 6.5 [3.8 to 9.2] | 6.3 [6 to 6.6]
  Bodily pain | 19.8 [13.2 to 26.4] | 3.9 [0.5 to 7.3] | 1.8 [1 to 4.6]
  General health | 13 [6.4 to 19.6] | 9.7 [8.2 to 11.2] | 11.6 [9.1 to 14.1]
  Vitality | 7.2 [5 to 9.4] | 3.9 [2.2 to 5.6] | 6.5 [4.9 to 8.1]
  Social functioning | 18.4 [9.2 to 27.6] | 10.4 [5.2 to 15.6] | 8.2 [5.3 to 11.1]
  Role emotional | 30.4 [17.9 to 42.9] | 12.8 [5.5 to 18.5] | 11.4 [8.5 to 14.3]
  Mental health | 14.4 [8.3 to 20.5] | 8.7 [5.6 to 11.8] | 11 [6.3 to 15.7]

2. Primary Outcome: Changes in the Quality of Life During the Treatment (Visit V0 vs Visit V3) Based on Results of All Groups of Patients
Description: QoL assessment using the SF36 scale questioner ( assessment of QoL quastions) - added to the Referance The Short Form (36) Health Survey (SF36 ) scale questioner was used. SF36 is is a 36-item, patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Time Frame: 1 month after presenting to a doctor
Measure: Mean (Full Range); unit: units on a scale
Groups:
- All Patients Suffering From Acute or Chronic Hemorrhoids Within 1 Month After Presenting to a Doctor: All groups of patients suffering from acute or chronic hemorrhoids within 1 month after presenting to a doctor (medical therapy, minimally invasive procedures, and surgical interventions)
Arm/Group | All Patients Suffering From Acute or Chronic Hemorrhoids Within 1 Month After Presenting to a Doctor
Number analyzed (Participants) | 1032
units on a scale
  Physical functioning | 13.8 [5.6 to 22]
  Role physical | 9.2 [7.6 to 10.8]
  Bodily pain | 8.8 [5.4 to 12.2]
  General health | 11.5 [8.9 to 14.1]
  Vitality | 6 [4.1 to 7.9]
  Social functioning | 12 [6.8 to 17.2]
  Mental health | 11.4 [6.7 to 16.1]
  Role emotional | 17.5 [11.4 to 23.6]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Conservative Treatment of Hemmorhoid | Combined Treatment of Hemmorhoid | Surgical Treatment of Hemmorhoid
All-Cause Mortality (participants affected / at risk) | 0/311 | 0/298 | 0/423
Serious Adverse Events (participants affected / at risk) | 0/311 | 0/298 | 1/423
Other Adverse Events (participants affected / at risk) | 0/311 | 0/298 | 0/423
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conservative Treatment of Hemmorhoid (N=311) | Combined Treatment of Hemmorhoid (N=298) | Surgical Treatment of Hemmorhoid (N=423)
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 (1) — Diarrhea was considered as serious (medically significant) as it resulted in worsening of post-operative healing and increase of pain syndrome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT03743311/Prot_SAP_000.pdf
  • Informed Consent Form (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT03743311/ICF_001.pdf